CLINICAL TRIAL: NCT06455514
Title: Neuroprotection Following Cardiac Arrest: A Randomized Control Trial of Magnesium
Brief Title: Post-CA Neuroprotection With Magnesium
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20-00262; 1R34HL166859-01A1 (NIH)
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Arrest; Return of Spontaneous Circulation
MeSH Terms: conditions — Heart Arrest | interventions — Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Magnesium Sulfate (Experimental): Treatment of initial magnesium sulfate bolus followed by a continuous drip.
  Interventions: Drug: Magnesium Sulfate
- Saline solution (Placebo Comparator): Treatment of equivalent volume of normal saline.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Magnesium Sulfate — 4 g of magnesium sulfate intravenously within 2 hours of Return of Spontaneous Circulation (ROSC), followed by a continuous drip (16 g) over 24 hours
  Arms: Magnesium Sulfate
Drug: Saline — Control subjects will receive an equivalent volume of normal saline intravenously.
  Arms: Saline solution

SUMMARY:
The purpose of this pilot interventional study is to collect preliminary data on administering magnesium sulfate as a neuroprotective medication in patients who achieved Return of Spontaneous Circulation (ROSC) following Cardiac Arrest (CA). The primary aims are to assess the feasibility and safety of administering magnesium and measure serum markers of neuronal injury at prespecified time points in the post-cardiac arrest period. Because this is a pilot study with a limited sample size, the primary objective is to evaluate the precision and stability of the collected measures to inform the design and formal analysis in a larger trial.

ELIGIBILITY:
Inclusion Criteria:

* Documented post-cardiac arrest patient with Return of Spontaneous Circulation (ROSC) achieved <2 hours prior to recruitment

Exclusion Criteria:

* Age < 18 years or > 85 years
* Traumatic cardiac arrests
* Unsustained ROSC (<20 minutes)
* Patient who is responsive/able to follow motor commands within 1 hour of achieving ROSC
* Plan for withdrawal of life support within 72 hours of ROSC
* Known pregnant women at the time of the cardiac arrest
* Known prisoners at the time of the cardiac arrest
* Subjects who have a medical o social condition that would make them inappropriate for the study based on the PI's or clinical team judgement.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of cases where successful randomization occurred | Through study completion, an average of 90 days
Proportion of cases where Magnesium (Mg) or saline bolus was delivered with a goal of <2 h after return of spontaneous circulation (ROSC) | Through study completion, an average of 90 days
Proportion of cases with adherence to treatment protocol | Through study completion, an average of 90 days
  Assessment of adherence will involve reviewing chart data to evaluate the timing of medication order placement and timing of administration by the nurse.
Proportion of cases for which serum is successfully drawn and analyzed | Through study completion, an average of 90 days
Proportion of cases where patient's Cerebral Performance Category Score (CPC) status is assessed | At hospital discharge, on average 3 weeks
  The CPC assessment score will be derived from the patient's electronic medical record (EMR).
Proportion of cases where patient's CPC status is assessed | Day 30
  The CPC assessment score will be derived from the patient's EMR.
Proportion of cases where patient's CPC status is assessed | Day 90
  The CPC assessment score will be derived from the patient's EMR.

SECONDARY OUTCOMES:
Number of participants with adverse reactions related to magnesium therapy | Through study completion, an average of 90 days
Proportion of cases for which magnesium levels are found to be >6 mg/dl | Through study completion, an average of 90 days
Proportion of cases for which magnesium levels are found to be 8.1-10 mg/dl | Through study completion, an average of 90 days
Proportion of cases for which magnesium levels are found to be >10 mg/dl | Through study completion, an average of 90 days
All-cause mortality | Day 90
  Mortality due to all causes
Proportion of patients with unfavorable neurological outcomes | At hospital discharge, on average 3 weeks
  The Cerebral Performance Category (CPC) score is a five-point scale used to assess neurological outcome after cardiac arrest and other events. Scores range from 1 to 5, a score of 1 or 2 is considered a favorable outcome, and scores of 3, 4, or 5 are considered an unfavorable outcome (severe neurological disability, persistent vegetative state or death).
Proportion of patients with unfavorable neurological outcomes | Day 30
  The Cerebral Performance Category (CPC) score is a five-point scale used to assess neurological outcome after cardiac arrest and other events. Scores range from 1 to 5, a score of 1 or 2 is considered a favorable outcome, and scores of 3, 4, or 5 are considered an unfavorable outcome (severe neurological disability, persistent vegetative state or death).
Proportion of patients with unfavorable neurological outcomes | Day 90
  The Cerebral Performance Category (CPC) score is a five-point scale used to assess neurological outcome after cardiac arrest and other events. Scores range from 1 to 5, a score of 1 or 2 is considered a favorable outcome, and scores of 3, 4, or 5 are considered an unfavorable outcome (severe neurological disability, persistent vegetative state or death).

CONTACTS AND LOCATIONS:
Overall Officials: Sam Parnia, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Sam.Parnia@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data upon reasonable request. Requests should be directed to Sam.Parnia@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.